CLINICAL TRIAL: NCT06954155
Title: Tenecteplase Reperfusion Therapy in Acute Ischemic Cerebrovascular Events-BEYOND--A Multicenter, Prospective, Randomized, Open Label, Blinded-endpoint (PROBE) Controlled Trial of Tenecteplase Versus Standard Medical Treatment for Acute Ischemic Stroke Due to Large Vessel Occlusion With Perfusion Mismatch 24 to 72 Hours of Symptom Onset
Brief Title: Tenecteplase Reperfusion Therapy in Acute Ischemic Cerebrovascular Events-BEYOND
Acronym: TRACE-BEYOND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA2024YJ007
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: ischemic stroke; tenecteplase; beyond 24 hours
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (0.25 mg/kg) (Experimental): Tenecteplase (0.25 mg/kg, max 25 mg)
  Interventions: Drug: Tenecteplase (0.25mg/kg)
- Standard medical treatment (Active Comparator): Aspirin combined with clopidogrel, aspirin alone, or clopidogrel alone
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Drug: Tenecteplase (0.25mg/kg) — Each vial of tenecteplase is reconstituted with 3 ml sterile water for injection and adjusted to a concentration of 5.33 mg/ml. Calculate the total amount of drug according to the subject's actual body weight and measure the required drug volume. The maximum dose should not exceed 25mg. Tenecteplase should be given as a single, intravenous bolus (within 5-10 seconds).
  Arms: Tenecteplase (0.25 mg/kg)
Drug: Standard medical treatment — Aspirin combined with clopidogrel, aspirin alone, or clopidogrel alone after randomization at the discretion of site researchers according to Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023.
  Arms: Standard medical treatment

SUMMARY:
The benefit-risk profile of thrombolysis for acute ischemic strokes beyond 24 hours has never been investigated. We initiated a multicenter, prospective, randomized, open label, blinded-endpoint (PROBE) controlled trial to assess the safety and efficacy of tenecteplase (0.25mg/kg, max 25mg) versus standard medical treatment in acute ischemic stroke due to large vessel occlusion between 24-72 hours of symptom onset (including wake-up stroke and unwitnessed stroke).

DETAILED DESCRIPTION:
Adult acute ischemic stroke patients due to large vessel occlusion (Middle cerebral artery M1 or M2 occlusion confirmed by CTA/MRA) with baseline National Institutes of Health Stroke Scale (NIHSS) 6-25 will be enrolled in this trial. We use perfusion imaging to select subjects and the enrolled patients have target mismatch profile on CTP or MRI+PWI (ischemic core volume <70mL, mismatch ratio ≥1.8, and mismatch volume ≥15mL). We will randomly assign patients who have salvageable brain tissue as identified on perfusion imaging to receive tenecteplase (at a dose of 0.25 mg per kilogram of body weight; maximum dose, 25 mg) or standard medical treatment 24 to 72 hours after the time that the patient was last known to be well (including after stroke on awakening and unwitnessed stroke). The primary outcome is the proportion of patients with an mRS score ≤ 1 at 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Acute ischemic stroke symptom onset between 24 to 72 hours prior to enrollment; including wake-up stroke and unwitnessed stroke, onset time refers to 'last-seen normal time';
3. Pre-stroke modified Rankin scale (mRS) score ≤1;
4. Baseline National Institutes of Health Stroke Scale (NIHSS) 6-25 (both inclusive);
5. Neuroimaging:

   1. Middle cerebral artery M1 or M2 occlusion confirmed by CTA/MRA, middle cerebral artery M1 or M2 being responsible for signs and symptoms of acute ischemic stroke;
   2. target mismatch profile on CTP or MRI+PWI (ischemic core volume <70mL, mismatch ratio ≥1.8, and mismatch volume ≥15mL);
6. Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

1. Present as a significant low-density lesion on CT
2. Allergy to tenecteplase
3. Rapidly improving symptoms at the discretion of the investigator
4. NIHSS consciousness score 1a >2, or epileptic seizure, hemiplegia after seizures (Todd's palsy) or other neurological/mental illness such that the patient is not able to cooperate or unwilling to cooperate
5. Persistent blood pressure elevation (systolic ≥185 mmHg or diastolic ≥110 mmHg), despite blood pressure-lowering treatment
6. Blood glucose <2.8 or >22.2 mmol/L (point of care glucose testing is acceptable)
7. Active internal bleeding or at high risk of bleeding, e.g., major surgery, trauma or gastrointestinal or urinary tract hemorrhage within the previous 21 days, or arterial puncture at a non-compressible site within the previous 7 days
8. Any known impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, then INR >1.7 or prothrombin time >15 seconds; use of any direct thrombin inhibitors or direct factor Xa inhibitors during the last 48 hours unless reversal of effect can be achieved with a reversal agent; any full dose heparin/heparinoid during the last 24 hours or with an aPTT greater than the upper limit of normal
9. Known defect of platelet function or platelet count below 100,000/mm3 (NB patients taking antiplatelet medication can be included)
10. Ischemic stroke or myocardial infarction in previous 3 months, previous intracranial hemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm, arteriovenous malformation, or giant aneurysm
11. Any terminal illness such that the patient would not be expected to survive more than 1 year
12. Unable to perform CTP or PWI
13. Hypodensity in >1/3 MCA territory on non-contrast CT
14. Acute or past intracerebral hemorrhage (ICH) identified by CT or MRI
15. Multiple arterial occlusion (bilateral MCA occlusion, MCA occlusion accompanied with basilar occlusion)
16. Pregnant women, nursing mothers, or reluctance to use effective contraceptive measures during the period of trial
17. Unlikely to adhere to the trial protocol or follow-up
18. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study
19. Participation in other interventional clinical trials within the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
mRS score ≤ 1 at 90 days | 90 days
  The proportion of patients with an mRS score ≤ 1 at 90 days

SECONDARY OUTCOMES:
mRS score | 90 days
  Ordinal distribution of mRS at 90 days (shift analysis)
mRS score ≤ 2 at 90 days | 90 days
  The proportion of patients with an mRS score of 0-2
early neurological improvement at 24h after randomization | 24 hours
  The rate of early neurological improvement at 24h after randomization (defined as a NIHSS score ≤1 or ≥4 points compared with baseline)
improvement on reperfusion at 24h after randomization | 24 hours
  The rate of improvement on reperfusion at 24h after randomization (improved by 90% on Tmax > 6s)
complete recanalization at 24h after randomization | 24 hours
  The rate of complete recanalization at 24h after randomization (defined as an AOL score of 3)
Symptomatic intracranial hemorrhage within 36 hours | 36 hours
  Symptomatic intracranial hemorrhage within 36 hours (defined by the ECASS III criteria)
All-cause mortality at 90 days | 90 days
  All-cause mortality at 90 days
Systemic bleeding at 90 days | 90 days
  Systemic bleeding at 90 days (defined by the GUSTO criteria: moderate and severe bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing tiantan hospital, Beijing, China